CLINICAL TRIAL: NCT03157921
Title: Prevalence of Spontaneous Ovulation and Pregnancy in Patients With Polycystic Ovary Syndrome
Brief Title: Prevalence of Pregnancy in Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer of obstetrics and gynecology, Assiut University
Other Study IDs: 17100186
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: transvaginal ultrasound — assessment of ovarian volume and antral follicle count
Diagnostic Test: Hormonal levels — follicle stimulating hormone level, luteinizing hormone level and anti-mullerian hormone level

SUMMARY:
Polycystic ovary syndrome is the most common endocrine disorder in women of reproductive age, with a prevalence of approximately 5-10%. Polycystic ovary syndrome is diagnosed according to Rotterdam criteria by at least two of the following three key features: oligomenorrhea or amenorrhea; clinical and/or biochemical signs of hyperandrogenism; the presence of polycystic ovaries on ultrasound and exclusion of other endocrine disorders including hyperprolactinemia, thyroid dysfunction and congenital adrenal hyperplasia. Polycystic ovary syndrome is also associated with insulin resistance, obesity and disorders of lipid metabolism, as well as infertility, although these findings have not been addressed in the Rotterdam criteria. Polycystic ovary syndrome is the major cause of anovulatory infertility. The recent studies suggest that anovulation resulting from ovarian follicle abnormalities in Polycystic ovary syndrome patients are 2-fold of normal ovaries. Firstly, early follicular growth is excessive, thus women with Polycystic ovary syndrome are characterized by an excessive number of small antral follicles (2- to 3-fold of normal ovaries). Secondly, the selection of one follicle from the increased pool of selectable follicles and its further maturation to a dominant follicle does not occur. This second abnormality in the folliculogenesis can cause menstrual dysfunction presented as oligomenorrhea or amenorrhea. Historically, Polycystic ovary syndrome treatment has not been curative in nature, instead treatments focus on resolution of clinical manifestations of the disease.

ELIGIBILITY:
Inclusion Criteria:

* infertile women
* age from 18 to 40 years
* poly-cystic ovary syndrome
* Body mass index 18.5-35 kg/m2

Exclusion Criteria:

1. Endocrine disorders (cushing syndrome-congenital adrenal hyperplasia)
2. Systemic disease
3. Use of oral contraceptive,glucocorticoid and antiandrogen
4. Use of ovulation induction or dopaminergic agents
5. Use of antidiabetes, anti obesity drugs
6. history of tubal or ovarian surgery

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: infertile women with poly-cystic ovary syndrome
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of poly-cystic ovarian syndrome women who will be ovulated | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided